CLINICAL TRIAL: NCT06815445
Title: Postoperative Pain and Blood Loss of Non-use Compared to Partial-use of a Tourniquet in Bilateral Total Knee Replacement: A Randomized- Control Trial
Brief Title: Postoperative Pain and Blood Loss of Non-use Compared to Partial-use of a Tourniquet in Bilateral Total Knee Replacement
Acronym: TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 043/2566
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative; Total Knee Replacement; Tourniquet
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study divided into 2 groups. This study was designed to compare the effect of NTU vs BOO in the patients underwent bilateral TKA.
  It is a crossover design to compare each knee in each group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know whether which group are using tourniquet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-use of a tourniquet (NTU) (Experimental): No tourniquet is used throughout the surgery.
  Interventions: Procedure: None tourniquet
- Partial-use of a tourniquet (Active Comparator): Partial use of a tourniquet is throughout the surgery.
  Interventions: Procedure: None tourniquet

INTERVENTIONS:
Procedure: None tourniquet — No tourniquet is used throughout the surgery.

SUMMARY:
Postoperative pain and blood loss of non-use compared to partial-use of a tourniquet in bilateral total knee replacement: A Randomized- Control Trial This study aimed to compare the effects of non-use (NTU) and partial-use (before osteotomy to skin closure; BOO) of a tourniquet in bilateral total knee arthroplasty (TKA) on postoperative pain and complications.

DETAILED DESCRIPTION:
Despite numerous meta-analyses, and randomized-control trials (RCTs), there is still no conclusive evidence on the most effective, and efficient method of using a tourniquet.

There is gap of knowledge of method of tourniquet usage. Hence this study will provide the best method to apply tourniquet.

ELIGIBILITY:
Inclusion Criteria:

* patients with over 50 years of age and diagnosed with bilateral severe knee osteoarthritis undergoing bilateral TKA

Exclusion Criteria:

* patients having undergone previous knee surgery
* patients being subject to uncontrolled hypertension, coagulopathy, or recent knee sepsis
* patients with an ASA physical status grade > 2,
* inability to use patient-controlled analgesia (PCA), such as communication, or cognitive issues, or those patients who were allergic to medications used in the treatment process.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | At postoperative Day1,2,3,4
  Morphine consumption and Visual analog scale for pain minimum 0, maximum 10

SECONDARY OUTCOMES:
Blood loss | At postoperative Day1,2,3,4
  Pre operative hematocrit and post operative hematocrit change

CONTACTS AND LOCATIONS:
Overall Officials: Thada Wipatasinlapin, MD, Principal Investigator — Queen Savang Vadhana Memorial Hospital, Thailand
Locations (1):
- Thada Wipatasinlapin, Chon Buri, Sriracha, Thailand